CLINICAL TRIAL: NCT04781530
Title: ADEQUATE Advanced Diagnostics for Enhanced QUality of Antibiotic Prescription in Respiratory Tract Infections in Emergency Rooms - Paediatric
Brief Title: Advanced Diagnostics for Enhanced QUality of Antibiotic Prescription in Respiratory Tract Infections in Emergency Rooms
Acronym: ADEQUATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: BioMérieux (Industry); Universiteit Antwerpen (Other); St George's, University of London (Other); University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADEQUATE
Record Dates: First submitted 2021-02-02; First posted 2021-03-04 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-12

CONDITIONS: Community-acquired Acute Lower Respiratory Infection
Keywords: community-acquired pneumonia; point-of-care test; rapid diagnostics
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Masking Description: The trial is unblinded / open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Device) (Experimental): Diagnostic Test: BioFire
  A molecular rapid syndromic testing platform, using the following panel:
  BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus) In addition to standard of care
  Interventions: Device: BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus)
- Control (Standard of Care) (No Intervention): Standard of Care

INTERVENTIONS:
Device: BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus) — BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus): Nasopharyngeal swab
  Arms: Intervention (Device)

SUMMARY:
This study is a randomized controlled trial where participants are randomly assigned in a 1:1 ratio to either a rapid test group or a control group. Standard care is provided in the control group. Follow-up is conducted until discharge from the hospital, followed by telephone check-ins and completion of questionnaires by the participants themselves or their proxies until 30 days after randomization. Children of any age presenting at selected participating sites with acute respiratory tract infections, where initial treatment decisions are uncertain, are eligible to participate. The study aims to enrol 520 participants and involves Paediatric Emergency Rooms across Europe.

DETAILED DESCRIPTION:
Background. Community-acquired acute respiratory tract infections (CA-ARTI) are among the most frequent infectious diseases worldwide. Uncomplicated ARTI is the most frequent cause of inappropriate antibiotic use, and there is a need of more judicious antibiotic prescribing to prevent exposure to drug-related adverse events and selection of antibiotic resistance. There is a need to assess the impact of rapid syndromic diagnostic testing in patients with CA-ARTI presenting to Emergency Rooms on clinical decision making related to hospitalisation and prescription of antibiotics. At the same time it must be determined whether the decisions guided by the rapid syndromic diagnostic testing results do not compromise patient safety.

Trial objective: To assess the impact of rapid diagnostic testing in patients with ARTI at the emergency department, on (1) hospital admission rates, (2) antimicrobial prescriptions (days of treatment) and (3) non-inferiority in terms of clinical outcome.

Secondary objectives include health care utilisation, time away from school or routine childcare arrangements and quality of life.

In an ancillary study, changing patterns in microbiological colonisation of the oropharynx following different management strategies will be assessed in a subset of participants.

Study design: Individually randomised controlled trial, randomisation 1:1 to either a rapid test group (intervention described below) or a control group, with management according to standard of care at the local facility. Follow-up until discharge from hospital and thereafter by telephone follow-up and self (or proxy)-completion questionnaires until 30 days after randomisation.

Study population: Children of any age consulting in selected participating sites with CA-ARTI, in which there is initial uncertainty about treatment and management decisions, after provision of informed consent by parent(s) or legal guardian.

Study Intervention: The diagnostic intervention is rapid syndromic testing on a nasopharyngeal swab with BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus) (licensed for routine use at all trial sites), results expected within four hours from sample collection.

Co-primary endpoints:

Hierarchical nested analysis design of:

* Days alive out of hospital (superiority endpoint), within 14 days after study enrolment
* Days on Therapy (DOT) with antibiotics (superiority endpoint), within 14 days after study enrolment

Secondary endpoints Adverse outcome (non-inferiority safety endpoint)

•Safety endpoint: For initially hospitalised patients: i) any readmission, ii) ICU admission => 24 hours after hospitalisation, or iii) death, within 30 days after study enrolment

For initially non-admitted patients: any admission or death within 30 days after study enrolment.

* Direct costs and indirect costs within 30 days after enrolment.
* Change in quality of life as determined by EQ-5D-5L (or suitable alternative for age), days away from usual childcare routine or school and healthcare utilisation on day 1, 14, and 30 after enrolment.
* Microbiological results obtained as standard of care and with the diagnostic intervention
* Empirical antibiotics, antibiotic type switches, de-escalation based on antimicrobial agent categories. Prescription of antivirals during the main study.
* Detection of antimicrobial resistance (carriage or infection) related to the diagnostic intervention results compared to standard of care and impact on antimicrobial stewardship guidelines and prevention of hospital acquired infections.
* Impact on decisions regarding isolation measures related to test result.

ELIGIBILITY:
Inclusion Criteria:

1. Children of any age presenting to the Emergency Room with an acute illness (present for 14 days or less) with Temperature ≥38.0°C measured at presentation or reported within the previous 24 hours

   AND at least two of the below:
   * Cough
   * Abnormal sounds on chest auscultation (crackles, reduced breath sounds, bronchial breathing, wheezing)
   * Clinical signs of dyspnea (chest indrawing, nasal flaring, grunting)
   * Signs of respiratory dysfunction: tachypnoea for age or decreased oxygen saturation (<92% in room air)
   * Signs of reduced general state: poor feeding, vomiting or lethargy/drowsiness
2. At time of screening:

   * Patient has undergone first assessment by managing clinical team (doctor or nurse, incl. triage)
   * Hospitalisation is not yet determined, i.e. neither by clinical presentation definitely requiring hospitalisation (e.g. per local guideline) nor by fixed decision of managing clinical team; admission to a short-stay unit or surveillance unit is not considered a hospitalisation for this trial
   * Antibiotic treatment or hospitalisation is being considered
   * The rapid syndromic diagnostic test result can be awaited for up to 4 hours before the decision to discharge the patient or to initiate antibiotic treatment is made

Exclusion Criteria:

1. Development of ARTI more than 48 hours after hospital admission (hospital acquired);
2. Patients with a severe underlying medical condition dictating management decisions including hospitalisation and/or antibiotic treatment (e.g cystic fibrosis, immunosuppression);
3. Less than 14 days since the last episode of respiratory tract infection;
4. Confirmed pregnancy and/or breastfeeding;
5. Any clinically significant abnormality identified at the time of screening that in the judgment of the Investigator would preclude safe completion of the study or constrain endpoints assessment such as major systemic diseases or patients with short life expectancy;
6. Inability to obtain informed consent;
7. Alternative noninfectious diagnosis that explains clinical symptoms.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 522 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Days alive out of hospital (superiority endpoint), within 14 days after study enrolment | 14 days
  Days alive out of hospital (superiority endpoint), within 14 days after study enrolment
Days on Therapy (DOT) with antibiotics (superiority endpoint), within 14 days after study enrolment | 14 days
  Days on Therapy (DOT) with antibiotics (superiority endpoint), within 14 days after study enrolment
Adverse outcome (non-inferiority safety endpoint) | 30 days
  Adverse outcome (non-inferiority safety endpoint)
  * For initially non-admitted patients: any admission or death within 30 days
  * For initially hospitalised patients: i) any readmission, ii) ICU admission >= 24 hours after hospitalisation, or iii) death, all within 30 days

SECONDARY OUTCOMES:
Direct costs and indirect costs within 30 days after enrolment. | 30 days
  * Cost of healthcare within 30 days after enrolment, including hospital and ICU days, utilisation of non-hospital services and cost of anti-infective and concomitant medication
  * Cost of workdays lost within 30 days, including days for childcare
Quality of life as determined by EQ5D-5L (or suitable alternative for age), days away from usual childcare routine or school and healthcare utilisation on day 1, 14, and 30 after enrolment. | 1, 14 and 30 days
  Quality of life as determined by EQ5D-5L (or suitable alternative for age), days away from usual childcare routine or school and healthcare utilisation on day 1, 14, and 30 after enrolment.
Microbiological results obtained as standard of care and with the diagnostic intervention | Day 1
  Proportion of participants with an identified respiratory pathogen in both study groups on randomisation day samples.
Empirical antibiotics based on antimicrobial agent categories | Day 1 - Day 14
  Proportion of participants on non-first-line anti-infective regimens (as defined by local guidelines)
Antibiotic type switches and de-escalation based on antimicrobial agent categories | Day 1 - Day 14
  Time to de-escalation and time to stop of anti-infective therapy
Detection of antimicrobial resistance (carriage or infection) related to the diagnostic intervention results compared to standard of care and impact on antimicrobial stewardship guidelines and prevention of hospital acquired infections | >7 days after randomisation
  Proportion of hospitalised participants with detection of cephalosporin-, carbapenem- or chinolone-resistant Enterobacteriaceae on any standard of care samples >7 days after randomisation
Impact on decisions regarding isolation measures related to test result. | Day 1 - Day 30
  Hours in individual or cohort isolation in hospitalised participants

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bielicki, PhD, Principal Investigator — St George's, University of London
Locations (6):
- University Children's Hospital Tuebingen, Tübingen, Germany
- Hippokration Hospital of Thessaloniki, Thessaloniki, Greece
- Hospital Universitario 12 de Octubre, Spain, Madrid, Spain
- Switzerland (2):
  - University Children's Hospital Basel (UKBB), Basel, Canton of Basel-City
  - Ospedale Regionale Bellinzona e Valli, Bellinzona
- University Hospital of Lewisham, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] ADEQUATE Paediatric Trial Group. Randomised multicentre effectiveness trial of rapid syndromic testing by panel assay in children presenting to European emergency departments with acute respiratory infections-trial protocol for the ADEQUATE Paediatric trial. BMJ Open. 2024 Apr 25;14(4):e076338. doi: 10.1136/bmjopen-2023-076338. PMID 38670622

DOCUMENTS (2):
  • Study Protocol (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT04781530/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT04781530/SAP_003.pdf